CLINICAL TRIAL: NCT00006258
Title: Dose Intensive Chemotherapy for Patients Greater Than or Equal To 10 Years of Age With Newly Diagnosed High Stage Medulloblastoma, Supratentorial Primitive Neuroectodermal Tumors (PNET) and Ependymoma: A Feasibility Study of an Intensive Induction Chemotherapy Regimen Followed by Standard Irradiation
Brief Title: Combination Chemotherapy Followed by Radiation Therapy in Treating Patients With Medulloblastoma, Supratentorial Primitive Neuroectodermal Tumor, or Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CHLA-NYU-0002H; CDR0000068192 (Registry Identifier: PDQ (Physician Data Query)); NYU-0027H; NCI-G00-1852
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2004-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; adult medulloblastoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult ependymoblastoma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma; newly diagnosed childhood ependymoma; adult supratentorial primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Central Nervous System Neoplasms; Medulloblastoma; Ependymoma; Neuroectodermal Tumors, Primitive | interventions — Filgrastim; Cisplatin; Cyclophosphamide; Etoposide; Methotrexate; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: methotrexate
Drug: vincristine sulfate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug or combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by radiation therapy in treating patients who have surgically resected, newly diagnosed medulloblastoma or supratentorial primitive neuroectodermal tumor, or incompletely resected ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of adjuvant dose-intensive induction chemotherapy with cisplatin, vincristine, cyclophosphamide, and etoposide with or without methotrexate followed by standard radiotherapy in patients with surgically resected, newly diagnosed high stage medulloblastoma or supratentorial primitive neuroectodermal tumor, or incompletely resected ependymoma.
* Determine the response rate, time to progression, overall survival, and pattern of failure in these patients treated with this regimen.

OUTLINE: Patients receive dose-intensive induction chemotherapy consisting of cisplatin IV over 6 hours on day 0; vincristine IV on days 0, 7, and 14; and etoposide and cyclophosphamide IV over 1 hour on days 1 and 2. Patients with M1+ disease (i.e., evidence of dissemination beyond primary tumor site) also receive methotrexate IV over 4 hours on day 3. Patients receive filgrastim (G-CSF) subcutaneously daily beginning on day 7 and continuing until blood counts recover. Chemotherapy continues every 21-28 days for a total of 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo radiotherapy 5 days a week for 6.5 weeks beginning 3-6 weeks after completion of chemotherapy.

Patients are followed at 6 weeks, then every 3 months for 2 years, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 6-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological confirmation of one of the following:

  * High stage medulloblastoma with neuraxis dissemination (Chang stage M1 or greater)
  * Primitive neuroectodermal tumor
  * Ependymoma

    * Incompletely resected on postoperative MRI or neurosurgical report
* Definitive prior surgery within 42 days of study

PATIENT CHARACTERISTICS:

Age:

* 10 to 65

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGPT less than 2.5 times upper limit of normal

Renal:

* Creatinine clearance greater than 60 mL/min

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior corticosteroids allowed
* No concurrent corticosteroids as antiemetics

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-11; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Finlay, MB, ChB, Study Chair — Children's Hospital Los Angeles
Locations (3):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Geisinger Medical Center, Danville, Pennsylvania
- Tom Baker Cancer Centre - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Dhodapkar K, Dunkel IJ, Gardner S, Sapp M, Thoron L, Finlay J. Preliminary results of dose intensive pre-irradiation chemotherapy in patients older than 10 years of age with high risk medulloblastoma and supratentorial primitive neuroectodermal tumors. Med Pediatr Oncol. 2002 Jan;38(1):47-8. doi: 10.1002/mpo.1262. No abstract available. PMID 11835236